CLINICAL TRIAL: NCT03503786
Title: MITO END-3: A Randomized Phase II Trial of Carboplatin+Paclitaxel Compared to Carboplatin+Paclitaxel+Avelumab in Advanced (Stage III-IV) or Recurrent Endometrial Cancer
Brief Title: Carboplatin, Paclitaxel With or Without Avelumab in Advanced or Recurrent Endometrial Cancer
Acronym: MITO END-3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO END-3; 2016-004403-31 (EudraCT Number)
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Cancer
Keywords: PD-L1 Expression; advanced endometrial cancer; recurrent endometrial cancer; Patient reported outcomes
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel; avelumab

STUDY DESIGN:
Intervention Model Description: Phase 2 randomized with a safety run-in cohort for the experimental arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): Carboplatin AUC 5+Paclitaxel 175 mg/m2 q 21days for 6-8 cycles and Avelumab
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Chemotherapy and avelumab (Experimental): Carboplatin AUC 5+ Paclitaxel 175 mg/ m2+Avelumab 10 mg/kg q 21days for 6 -8 cycles + Avelumab 10 mg/kg every 14 days until disease progression or unacceptable toxicity
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Avelumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC 5 i.v. every 3 weeks for 6 - 8 cycles
Drug: Paclitaxel — Paclitaxel 175 mg/m2 i.v. every 3 weeks for 6-8 cycles
Drug: Avelumab — Avelumab 10 mg/kg every 3 weeks for 6-8 cycles + Avelumab 10 mg/kg every 14 days until disease progression or unacceptable toxicity
  Arms: Chemotherapy and avelumab

SUMMARY:
This study aims to evaluate the safety and activity of the Avelumab in combination with Carboplatin-Paclitaxel in advanced or recurrent endometrial cancer

ELIGIBILITY:
Inclusion Criteria:

1. Female aged at least 18 years on day of signing informed consent
2. ECOG Performance Status of 0-1
3. Patients with newly diagnosed or recurrent endometrial cancer FIGO stage III-IV and histologically-confirmed (any histology except sarcoma and carcinosarcoma)
4. Patients may have received adjuvant treatment (platinum-based cytotoxic chemotherapy and/or radiotherapy). Patients having received prior chemotherapy must have completed their treatment at least 6 months prior to registration for protocol therapy. Patients having received prior radiotherapy must have completed their treatment at least 28 days prior to registration for protocol therapy
5. Have measurable disease based on RECIST v1.1 criteria
6. Availability of tumor samples for biomarker analysis
7. Endometrial cancer will include all carcinomas, including endometrioid carcinoma, papillary serous carcinoma, clear cell carcinoma
8. Adequate hematological function defined by absolute neutrophil count (ANC) ≥ 1500 × mm3, platelet count ≥ 100,000 × mm3, and hemoglobin ≥ 9 g/dL (may have been transfused)
9. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN for all subjects (or ≤ 5 x ULN if liver metastases are present)
10. Adequate renal function defined by an estimated creatinine clearance ≥ 50 mL/min according to the Cockcroft-Gault formula or serum creatinine ≤ 1.5 ULN (for local institutional standard method)
11. Alkaline phosphatase < 1.5 x ULN for the institution (if > 1.5 x ULN, then alkaline phosphatase liver fraction must be < 1.5 ULN)
12. Be willing and able to provide written informed consent/assent for the trial
13. Females of childbearing potential must have a negative serum pregnancy test (serum hCG) at screening. Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥1 year
14. Highly effective contraception for females if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1 % per year). Highly effective contraception is required at least 28 days prior, throughout and for at least 60 days after Avelumab treatment

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Patients with brain metastases, except those meeting the following criteria:

   * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
   * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
   * patients must be either off steroids or on a stable or decreasing dose of <10mg daily prednisone (or equivalent)
3. Prior Anticancer treatment for advanced disease and/or prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. Previous hormonal therapy for advanced disease is allowed, but treatment must be discontinued at least 28 days prior to registration for protocol therapy
4. History of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
5. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
6. Prior organ transplantation, including allogeneic stem cell transplantation
7. Significant acute or chronic infections including, among others:

   * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
   * Positive test for hepatitis B surface antigen and / or confirmatory hepatitis C RNA (if anti-hepatitis C antibody tested positive)
   * Evidence of interstitial lung disease or active non-infectious pneumonitis.
   * Active infection requiring systemic therapy
   * Known history of active Tuberculosis Bacillus (TB)
8. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

   * Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
   * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
   * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
9. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable
10. Another primary malignancy within the past five years (except for non-melanoma skin cancer and cervical carcinoma in situ).
11. Concurrent treatment with immunosuppressive or investigational agents EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
12. Active cardiac disease, defined as:

    * Myocardial infarction or unstable angina pectoris within 6 months of the first date of study therapy,
    * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrio-ventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
    * New York Heart Association (NYHA) Class III or greater congestive heart failure, or left ventricular ejection fraction of < 40%.
13. Known alcohol or drug abuse
14. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
15. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
16. All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma) including recent or active suicidal ideation or behavior, which, in the opinion of the Investigator, may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 18 months from beginning of treatment

SECONDARY OUTCOMES:
overall survival | 3 years
number of patients with complete and partial responses | 18 months
worst grade toxicity per patient | evaluated every 3 weeks up to 2 years
  according to Common Toxicity Criteria for Adverse Events v. 4.03
changes in patient-reported outcome (PRO) scores of quality of life and endometrial cancer disease and treatment related symptoms from baseline | up to 2 years
  European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C-30 En-24C QOL questionnaire C-30 En-24
changes in patient-reported outcome (PRO) scores of symptomatic toxicities during treatment | up to 2 years
  PRO-CTCAE questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Gennaro Daniele, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (11):
- Italy (11):
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS San Raffaele, Milan
  - Istituto Nazionale Tumori, Milan
  - AOU Policlinico Federico II, Napoli
  - AOU Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Silvestrini, Perugia
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Universitario Gemelli Università Cattolica del Sacro Cuore, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pignata S, Scambia G, Schettino C, Arenare L, Pisano C, Lombardi D, De Giorgi U, Andreetta C, Cinieri S, De Angelis C, Priolo D, Casanova C, Rosati M, Greco F, Zafarana E, Schiavetto I, Mammoliti S, Cecere SC, Salutari V, Scalone S, Farolfi A, Di Napoli M, Lorusso D, Gargiulo P, Califano D, Russo D, Spina A, De Cecio R, Chiodini P, Perrone F; MITO investigators. Carboplatin and paclitaxel plus avelumab compared with carboplatin and paclitaxel in advanced or recurrent endometrial cancer (MITO END-3): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2023 Mar;24(3):286-296. doi: 10.1016/S1470-2045(23)00016-5. Epub 2023 Feb 14. PMID 37052965